CLINICAL TRIAL: NCT05665283
Title: A Randomized Open Label Crossover Single Dose Bioequivalency Study of Ensartinib Capsules in Healthy Volunteers Under Fasted Conditions
Brief Title: A Single Dose BE Study of X-396 in Healthy Volunteers Under Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xcovery Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: XCV-X396-ONC-103
Record Dates: First submitted 2022-10-21; First posted 2022-12-27 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Bioequivalency
Keywords: Bioequivalency; Phase I
MeSH Terms: interventions — ensartinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reference Standard Group (Active Comparator): In Period 1, 32 healthy volunteers will divided evenly and randomly assigned to receive 1 dose of 100 mg capsules from either the test product or reference product.
  In Period 2 the same patients in each cohort will cross over and receive 1 dose of the 100 mg from the other group. These healthy volunteers will receive 1 dose from each of the 100 mg capsules manufactured by both processes.
  Interventions: Drug: Ensartinib Hydrochloride
- Test Standard Group (Active Comparator): In Period 1, 32 healthy volunteers will divided evenly and randomly assigned to receive 1 dose of 100 mg capsules from either the test product or reference product.
  In Period 2 the same patients in each cohort will cross over and receive 1 dose of the 100 mg from the other group. These healthy volunteers will receive 1 dose from each of the 100 mg capsules manufactured by both processes.
  Interventions: Drug: Ensartinib Hydrochloride

INTERVENTIONS:
Drug: Ensartinib Hydrochloride — oral ALK inhibitor
  Other Names: X-396

SUMMARY:
This is an open-label, Phase I single dose 2-part, crossover bioequivalence study under fasted conditions. The trial is designed to evaluate the pharmacokinetic parameters between single doses of 100mg ensartinib capsules manufactured by two different processes.

DETAILED DESCRIPTION:
A Phase I, randomized, open-label single dose, 2-part, crossover bioequivalence study under fasted conditions to compare 100 mg capsules manufactured using the proposed commercial manufacturing process to the corresponding capsules which were utilized in the Phase III clinical study manufactured by a different process. A total of 32 healthy subjects were divided evenly and were randomized into 1 of the 2 treatment sequences (T-R or R-T) prior to Period 1 dosing. Subjects received the test product (100 mg ensartinib hydrochloride capsules manufactured with the registration stability process) or the reference product (100 mg ensartinib hydrochloride capsules utilized in the Phase 3 trial) according to their assigned treatment sequence.

The single dose crossover study will have a minimum washout period of 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Females of non-childbearing potential and males age 18~55 years. Female subjects must be of non-childbearing potential (according to Appendix A), and have a negative serum pregnancy test at screening and a negative urine pregnancy test at (each) admission to the clinical research center.
2. Male subjects with female partners of child-bearing potential must use two forms of acceptable contraception (according to Appendix A).
3. Male body weight ≥ 50.0 kg or female body weight ≥ 45.0 kg; BMI between 18.0-32.0 kg/m2.
4. Generally in good health, with no history of any (in the opinion of the Investigator) clinically significant, chronic or serious cardiovascular, hepatic, renal, respiratory, blood and lymphatic system, endocrine, immune, mental, neurological, gastrointestinal diseases. Additionally, no abnormalities of clinical significance in vital sign examination, physical examination, clinical laboratory tests (blood routine, urinalysis, blood biochemistry, drug test, nicotine test, etc.), and 12-lead ECG.
5. No plan for sperm or egg donation during screening and for the next 6 months.
6. Able to provide written, informed consent before initiation of any study related procedures, and is able, in the opinion of the Investigator, to comply with all the requirements of the study.
7. Able to swallow oral medication.
8. Able to communicate well with the investigator and understand and comply with all study requirements.

Exclusion Criteria:

1. History of allergies or hypersensitivity to any excipient (microcrystalline cellulose, stearic acid, hydroxypropyl methylcellulose, or tartrazine, (a dye used in the ensartinib 100 mg capsules) or aspirin, or history of allergies to two or more kinds of drugs or foods.
2. History of clinically significant, in the opinion of the investigator, dysphagia or history of any gastrointestinal diseases that may affect drug absorption.
3. Received surgery within 3 months of the first dose, a history or have plans for a surgery during the study, that might affect absorption, distribution, metabolism, and excretion of drugs (e.g., gastrectomy, cholecystectomy, or other gastrointestinal tract surgery, except appendectomy).
4. The presence of diseases with abnormal clinical manifestations that need to be excluded, in the opinion of the investigator, including but not limited to nervous, cardiovascular, blood and lymphatic system, immune, renal, hepatic, gastrointestinal, respiratory, metabolic and skeletal diseases.
5. Venipuncture intolerance or history of blood phobia and needle sickness.
6. Drug abuse within 3 months of the first dose.
7. Donated ≥200 mL of blood (blood components) or had massive blood loss, received blood transfusion or blood products within 3 months of the first dose.
8. Males who are planning a pregnancy with a partner or sperm donation in upcoming 6 months.
9. The use of potent CYP3A inhibitors or inducers (see Appendix C in the trial protocol for details) and potent P-gp inhibitors (verapamil, cyclosporine A, dexverapamil) within 2 weeks before first dose.
10. Received any prescription drug, over-the-counter drug, herbal drug or vitamins within 2 weeks of the first dose. An exception is made for incidental use of acetaminophen or an NSAID, which is allowed up to admission to the clinical research center.
11. Received any vaccine within 4 weeks of the first dose.
12. Excessive smoking (more than 5 cigarettes/day) within 3 months of the first dose, or disagreed on avoiding use of any tobacco products during the trial.
13. Excessive alcohol use (more than 14 units of alcohol per week) (1 unit of alcohol ≈ 360 mL of beer, 45 mL of liquor at 40% ABV, or 150 mL of wine) within 3 months of the first dose, or unwilling to quit alcohol during the trial.
14. Excessive tea, coffee and/or caffeinated beverages (more than 8 cups, 250 ml for each cup) every day within 3 months of the first dose (amount based on investigator opinion)
15. Consumption of excessive dragon fruit, mango, pomelo, lime, carambola, or food or beverage products prepared within 7 days of the first dose (amount based on investigator opinion).
16. Have a special diet requirement and cannot accept an uniform diet.
17. The presence of abnormal vital sign findings of clinical significance. Normal ranges for reference (including cutoffs): systolic blood pressure 90~139 mmHg, diastolic blood pressure 50-89 mmHg, pulse 40-100 beats/min, temperature (oral) 35.4-37.7 °C, and breathing 10-20 breaths/min at a sitting position. The specific results are comprehensively judged by the investigator.
18. Abnormal findings in any item of laboratory tests and auxiliary tests, which are of clinical significance at the investigator's discretion.
19. Subject has any history of human immunodeficiency virus (HIV) or immunodeficiency or known diagnosis of hepatitis B or C.
20. Subject has history or diagnosis of cancer with the exception of basal cell carcinoma treated more than 3 years prior to first dose and without a recurrence.
21. An alcohol level greater than 0.0 mg/100mL as indicated by an alcohol breath test (ABT) or drug abuse screening test (morphine, methamphetamine, ketamine, ecstasy, and cannabis) positive.
22. Between screening and (first) admission on day -1: Those who had diseases or took drugs ineligible for enrollment in the opinion of the investigator in this period; Those who ate methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, energy drinks) or grapefruit (juice) from 48 hours (2 days) prior to (first) admission.
23. Previous participation in this study or subjects that are deemed by the investigator as not appropriate for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Cmax | 14 Days
  Maximum observed concentration
AUC(0-t) | 14 Days
  Area under the concentration time curve from time 0 to time of the last quantifiable
AUC(0-∞) | 14 Days
  Area under the concentration time curve from time 0 to infinity

SECONDARY OUTCOMES:
tmax | 14 Days
  Time to reach maximum observed plasma concentration
t1/2 | 14 Days
  Apparent terminal elimination half life
lz | 14 Days
  Terminal Phase elimination rate constant

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Selvaggi, MD, Principal Investigator — Xcovery Holdings, Inc.
Locations (1):
- ICON - Early Development Services, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No